CLINICAL TRIAL: NCT05843409
Title: Mindfulness-based Stress Reduction or Usual Treatment for Treatment of Chronic Pain in an Italian Hospital
Brief Title: Mindfulness-based Stress Reduction (MBSR) for Reduction of Chronic Pain and Drug Therapie
Acronym: Chronicare
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale di Lecco (Other)
Responsible Party: Principal Investigator, Vincenzo Damico, Principal Investigator: Vincenzo Damico, Registered Nurse, Doctor of Philosophy, Department of Anesthesia and Critical Care, Azienda Socio Sanitaria Territoriale of Lecco, Azienda Socio Sanitaria Territoriale di Lecco
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Chronicare
Record Dates: First submitted 2023-04-12; First posted 2023-05-06 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Normal drug therapie or usual treatment
- Intervention (Experimental): Normal drug therapie or usual treatment with add Mindfulness-based stress reduction (MBSR)
  Interventions: Behavioral: Mindfulness-based stress reduction (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction (MBSR) — Mindfulness-based stress reduction may be associated with short-term effects on pain intensity and physical functioning. Patients will be randomized into 2 groups. The experimental group will receive MBSR sessions, with the frequency and duration specified in the study protocol. The sessions will be free and carried out by expert staff
  Arms: Intervention

SUMMARY:
Mindfulness-Based Cognitive Therapy (MBCT) combines ideas of traditional cognitive therapies with meditative practices aimed at cultivating mindfulness. Mindfulness-based stress reduction (MBSR) is considered one of the original mindfulness-based interventions. It has been modified to be offered virtually,which has been useful throughout the COVID pandemic, and more importantly, has served to inform other mindfulness approaches, such as trauma-focused therapy. The investigators want to assess the efficacy of MBSR in patients with Chronic Pain undergoing drug treatment.

DETAILED DESCRIPTION:
Mindfulness helps develop the ability to observe and detach from our mental, sensory, and emotional states, and thus increases our awareness and ability to manage emotions.

In the experimental arm, some have been foreseen group sessions, in which a maximum of ten people participate on the Mindfulness-based stress reduction (MBSR).

The protocol provides for eight meetings (one and a half or two hours each) on a monthly basis, for a total duration, therefore, of twelve months.

ELIGIBILITY:
Inclusion Criteria:

* Patients being treated for Chronic Pain
* Patients with Chronic Pain in Pharmacological Therapy

Exclusion Criteria:

* Patients with Chronic Pain not in Pharmacological Therapy
* Patients without Chronic Pain

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Chronic pain assessed with the Brief Pain Inventory (BPI) | 1 year
  Chronic or persistent pain is pain that carries on for longer than 12 weeks despite medication or treatment.

SECONDARY OUTCOMES:
Quality of life assessore with EQ5D | 1 year
  Perceived quality of life in the 5 dimension of EQ5D
Drug assumption | 1 year
  Drug or therapy assumption by the patient for pain treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Damico, Principal Investigator — Rn PhD, Department of Anesthesia and Critical Care, Asst Lecco
Locations (1):
- ASST Lecco, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Damico V, Milani M, Murano L. Effect of Mindfulness-Based Stress Reduction on Patients With Chronic Pain: A Randomized Controlled Trial. Pain Manag Nurs. 2025 Oct;26(5):510-522. doi: 10.1016/j.pmn.2025.02.010. Epub 2025 Mar 13. PMID 40082096